CLINICAL TRIAL: NCT03561623
Title: Quantitative Spinal Cord Gray Matter Imaging in Post Polio Syndrome
Brief Title: Spinal Cord Gray Matter Imaging in Post Polio Syndrome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Other Study IDs: PPS_Cord
Record Dates: First submitted 2018-06-05; First posted 2018-06-19 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Post-polio Syndrome
MeSH Terms: conditions — Postpoliomyelitis Syndrome | interventions — Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Post Polio Syndrome: Post Polio syndrome diagnosed according to March of Dimes Criteria; 'magnetic resonance (MR) Imaging' will be performed including a 'quantitative muscle force assessment'
  Interventions: Other: magnetic resonance (MR) Imaging; Other: quantitative muscle force assessment
- Healthy controls: subjects age- and sex-matched; 'magnetic resonance (MR) Imaging' will be performed including a 'quantitative muscle force assessment'
  Interventions: Other: magnetic resonance (MR) Imaging; Other: quantitative muscle force assessment

INTERVENTIONS:
Other: magnetic resonance (MR) Imaging — MRI of spinal cord and brain
Other: quantitative muscle force assessment — quantitative assessment of muscle force

SUMMARY:
This is a longitudinal, observational study with the aims of comparing spinal cord gray matter areas in patients with Post-Polio Syndrome to age and sex matched healthy control subjects and to correlate atrophy with metrics of clinical disability.

DETAILED DESCRIPTION:
Post-Polio syndrome (PPS) is characterised by new muscle weakness, pain, and fatigue several years to decades after the acute polio infection. Pathomechanisms are not yet fully understood.

This is a longitudinal, observational study. The aims are (a) to detect spinal cord gray (and possibly) white matter atrophy in patients with Post Polio Syndrome in comparison to healthy age and sex matched control subjects both cross-sectionally and longitudinally and (b) to correlate spinal cord gray and white matter atrophy to metrics of clinical disability.

Investigators will assess 20 patients with Post-Polio syndrome and 20 control subjects at baseline and 48 weeks by MRI and clinically including quantitative muscle strength assessments.

ELIGIBILITY:
Inclusion Criteria:

* Prior paralytic poliomyelitis with evidence of motor neuron loss. This is confirmed by history of the acute paralytic illness, signs of residual weakness and atrophy of muscles on neuromuscular examination, and signs of motor neuron loss.
* a period of partial or complete functional recovery after acute paralytic poliomyelitis, followed by an interval (usually 15 years or more) of stable neuromuscular function.
* slowly progressive and persistent new muscle weakness or decreased endurance, with or without generalized fatigue, muscle atrophy, or muscle and joint pain. Symptoms that persist for at least a year.
* Exclusion of other neuromuscular, medical, and skeletal abnormalities as causes of symptoms.
* Patients older than 18 years at time of screening
* Ambulant
* Ability to walk 150 m in the 6 min walking distance (6MWT) with or without one or two walking sticks.

Exclusion Criteria:

* Previous (3 months or less) or concomitant participation in any other therapeutic trial
* known or suspected malignancy
* Other chronic disease or clinical relevant limitation of renal, liver, heart function according to discretion of investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 patients with Post-Polio Syndrome and 20 healthy age and sex matched control subjects were included in this study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
spinal cord gray matter (GM) area measured by MRI | change between baseline and year 1
  Change in spinal cord cross-sectional gray matter area measured at baseline and at year 1

SECONDARY OUTCOMES:
spinal cord white matter (WM) area measured by MRI | at baseline
  spinal cord cross-sectional white matter area
change in spinal cord white matter (WM) area measured by MRI | between baseline and year 1
  Change spinal cord cross-sectional white matter area
total spinal cord area measured by MRI | at baseline
  spinal cord total cross-sectional area
Change in total spinal cord area measured by MRI | between baseline and year 1
  Change in spinal cord total cross-sectional area
quantitative muscle strength measured by hand-held dynamometer | at baseline
  assessed by hand-held dynamometer
change in quantitative muscle strength measured by hand-held dynamometer | between baseline and year 1
  assessed by hand-held dynamometer
motor cortical thickness measured by MRI | at baseline
  motor cortical thickness
Change in motor cortical thickness measured by MRI | between baseline and year 1
  Change in motor cortical thickness

CONTACTS AND LOCATIONS:
Overall Officials: Regina Schlaeger, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Children's Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No